CLINICAL TRIAL: NCT05213481
Title: Phase I, Open-Label, Single-sequence, Cross-Over Study of the Effect of Multiple Doses of Carbamazepine on Single-Dose Tepotinib Pharmacokinetics in Healthy Participants
Brief Title: Tepotinib Drug-Drug Interaction Study With Carbamazepine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS200095_0051; 2021-003546-20 (EudraCT Number)
Record Dates: First submitted 2021-11-22; First posted 2022-01-28 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Healthy
Keywords: Clinical pharmacology; Metabolite; Induction of metabolism
MeSH Terms: interventions — tepotinib; Carbamazepine

STUDY DESIGN:
Intervention Model Description: This is a single sequence cross-over trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tepotinib then Carbamazepine (Experimental): Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 1 and Day 26 in the morning under fed state followed by Carbamazepine 100, 200 or 300mg oral dose under fed state twice daily at the same time each day in the morning and evening from Days 8 to Day 32
  Interventions: Drug: Tepotinib; Drug: Carbamazepine

INTERVENTIONS:
Drug: Tepotinib — Participants received Tepotinib hydrochloride hydrate film-coated tablet once daily with food on Day 1 and Day 26 in the morning.
Drug: Carbamazepine — Carbamazepine 100 mg twice daily at Day 8 and 9, 200 mg twice daily at Day 10 and 11, 300 mg twice daily from Day 12 to 32.

SUMMARY:
The purpose of this study was to assess the effect of multiple doses of carbamazepine on single- dose tepotinib pharmacokinetics in healthy participants. Study details include: Study Duration: up to about 10 weeks; Treatment Duration: single dose of tepotinib on Days 1 and 26, 25 days of treatment with carbamazepine (Days 8 to 32); Visit Frequency: residence in the Clinical Research Unit from Days -1 to 4 and Days 25 to 29, ambulatory daily visits from Days 5 to 24 and 30 to 33, and one ambulatory visit on Day 39.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy participants as determined by medical evaluation, including no clinically significant abnormality identified by medical history, cardiac monitoring, physical examination or laboratory evaluation and no active clinically significant disorder, condition, infection or disease that would pose a risk to participant safety or interfere with the study evaluation, procedures, or completion at Screening and Day -1
* Had a body weight within 50 and 100 kilogram (inclusive) and Body Mass Index (BMI) within the range greater than or equal (>=) 18.5 and less than or equal to (<=) 29.9 kilogram per meter square (inclusive) at Screening
* Male or female (not a Women of childbearing potential [WOCBP]). The Investigator confirms that each participant agrees to use appropriate contraception and barriers, if applicable. The contraception, barrier, and pregnancy testing requirements are below:
* Contraceptive use was consistent with local regulations on contraception methods for those participating in clinical studies. Male Participants: Agree to the following during the study intervention period and for at least 1 week after the last dose of study intervention: Refrain from donating fresh and unwashed sperm PLUS (+), either: Abstain from intercourse with a WOCBP.OR Use a male condom: When having sexual intercourse with a WOCBP, who is not currently pregnant, and instruct her to use a highly effective contraceptive method with a failure rate of < 1percent (%) per year
* Since a condom may break or leak. Not a WOCBP, confirmed at Screening, by fulfilling at least 1 of the following criteria: Females who are postmenopausal (age-related amenorrhea >= 12 consecutive months and increased Follicle-stimulating hormone (FSH)
* Documentation of irreversible surgical sterilization by hysterectomy, or bilateral oophorectomy, or bilateral salpingectomy
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History or presence of clinically relevant respiratory, gastrointestinal, renal, hepatic, hematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, connective tissue diseases or disorders, as determined by medical evaluation
* Participants with gall bladder removal or other relevant surgery of gastrointestinal tract (appendectomy is not considered as relevant)
* History of any malignancy except for adequately treated superficial basal cell carcinoma
* History of epilepsy
* Ascertained or presumptive allergy/hypersensitivity to the active drug substance and/or excipients; history of anaphylaxis to drugs or serious allergic reactions leading to hospitalization or any other allergy reaction in general, which the Investigator considers may affect the safety of the participant and/or outcome of the study
* Any condition, including findings in the laboratory tests, medical history, or other Screening assessments, that in the opinion of the Investigator constitutes an inappropriate risk or a contraindication for participation in the study or that could interfere with the study's objectives, conduct, or evaluation
* Use of any prescribed medicine or over-the-counter drug or dietary supplement, including herbal remedies, vitamins, and minerals, antacids and dietary supplements such as fish oils within 2 weeks or 5 times the half-life of the respective drug, whichever is longer, prior to the first administration of study intervention
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany, will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.merckgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0051
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 29 participants were screened, out of which 18 participants received the study drug.
Groups:
- Tepotinib Then Carbamazepine: Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 1 and Day 26 in the morning under fed state followed by Carbamazepine 100 mg twice daily at Day 8 and 9, 200 mg twice daily at Day 10 and 11, 300 mg twice daily from Day 12 to 32.
Period: Overall Study
Arm/Group | Tepotinib Then Carbamazepine
Started | 18
Completed | 14
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 00
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Tepotinib
Description: The AUC from time zero (= dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda (λ)z determination.
Time Frame: Predose 60 minutes before tepotinib dosing and 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 30, 38, 48, 60, 72, 96, 120, 144, and 168 hours post dose. Predose 60 minutes before carbamazepine dosing and 1, 1.5, 2, 3, 4, 6, and 8 hours post dose
Population: PK analysis set included all participants who had administered any dose of any study intervention and completed the study without any relevant protocol deviations and factors likely to affect the comparability of PK results. Here 'Overall number of participants analyzed' = overall number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours* nanograms per milliliter(h*ng/mL)
Groups:
- Tepotinib: Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 1.
- Tepotinib Then Carbamazepine: Participants received a single oral dose of Tepotinib 500 milligrams (mg) on Day 26 under fed state followed by Carbamazepine, 300 mg twice daily from Day 26 to 32.
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
hours* nanograms per milliliter(h*ng/mL) | 25101 (20.2) | 16738 (14.1)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve (AUC) From Time Zero to Time of Last Measurable Concentration (AUC0-tlast) of Tepotinib
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
h*ng/mL | 24069 (20.2) | 16272 (13.4)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per mililiter (ng/mL)
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
nanogram per mililiter (ng/mL) | 414 (15.4) | 372 (18.2)

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAES With Severity of Grade Greater or Equal to 3
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a study intervention. A serious adverse event (SAE) was any untoward medical occurrence that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAE's were those events with onset dates on or after the first administration of study intervention. Severity of abnormalities were evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) version [24.1].
  grade 1 : mild grade 2 : moderate grade 3 : severe or medically significant but not immediately life-threatening grade 4 : life threatening or disabling grade 5 : death related to AE
Time Frame: Baseline (Day 1) up to 10 Weeks
Population: Safety Analysis Set included all participants, who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 18
Participants
  Any TEAE | 17
  Any serious TEAE | 0
  Any TEAE of Grade ≥ 3 (severe) | 0

5. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Laboratory Values
Description: Number of participants with clinically significant change from baseline in laboratory parameters were reported. Clinical Significance was decided by the investigator. Laboratory investigation included hematology, biochemistry, urinalysis, and coagulation.
Time Frame: Baseline (Day 1) up to 10 Weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 18
Participants
  Hematology | 0
  Biochemistry | 0
  Urinalysis | 0
  Coagulation | 0

6. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Electrocardiogram (ECG)
Description: Number of participants with clinically significant change from baseline in ECG parameters were reported. Clinical Significance was decided by the investigator. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), Respiratory Rate, Pulse Rate, QRS, QT and QTcB calculated by the Bazett formula.
Time Frame: Baseline (Day 1) up to 10 Weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 18
Participants | 0

7. Secondary Outcome: Number of Participants With Clinically Meaningful Change From Baseline in Vital Signs
Description: Number of participants with clinically significant change from baseline in vital signs. Clinical Significance was decided by the investigator. Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate.
Time Frame: Baseline (Day 1) up to 10 Weeks
Population: The safety analysis set included all participants who had received any dose of the study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 18
Participants | 0

8. Secondary Outcome: Total Body Clearance of Drug From Plasma (CL/f) for Tepotinib
Description: CL/f following oral administration was calculated as Dose/AUC0-inf, where AUC0-inf calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastcalc/λz, where Clastcalc was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and λz was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
liter/hour | 17.9 (20.2) | 26.9 (14.1)

9. Secondary Outcome: Apparent Volume of Distribution (Vz/f) for Tepotinib
Description: Vz/F was defined as the apparent volume of distribution during the terminal phase following extravascular administration.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
liters | 801 (24.3) | 1157 (21.2)

10. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib
Description: The time to reach the maximum observed plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
Hours | 8.02 [3.0 to 16.0] | 8.0 [6.0 to 16.0]

11. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Tepotinib in Plasma
Description: t1/2 was defined as the time taken for the plasma concentration or the amount of drug in the body to be reduced by half.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Tepotinib | Tepotinib Then Carbamazepine
Number analyzed (Participants) | 17 | 14
Hours | 31.0 (19.4) | 29.8 (25.8)

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to 10 Weeks
Groups:
- Tepotinib: Participants received 500 mg of Tepotinib hydrochloride hydrate film coated tablet once daily with food on Day 1.
- Carbamazepine: Carbamazepine 100 mg twice daily at Day 8 and 9, 200 mg twice daily at Day 10 and 11, 300 mg twice daily from Day 12 to 25.
Arm/Group | Tepotinib | Carbamazepine | Tepotinib Then Carbamazepine
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 7/18 | 13/14 | 7/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tepotinib (N=18) | Carbamazepine (N=14) | Tepotinib Then Carbamazepine (N=14)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 1
Feeling drunk (General disorders) | 0 | 4 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0
Headache (Nervous system disorders) | 2 | 3 | 0
Hypersomnia (Nervous system disorders) | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hot flush (Vascular disorders) | 0 | 2 | 0
Diplopia (Eye disorders) | 0 | 2 | 0
Vision blurred (Eye disorders) | 0 | 2 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 3 | 1
Fatigue (General disorders) | 0 | 4 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 6 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abnormal faeces (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 0 | 0
Thirst (General disorders) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 3 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Head discomfort (Nervous system disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05213481/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT05213481/SAP_001.pdf